CLINICAL TRIAL: NCT02714478
Title: Efficacy of "Equistasi" on the Gait of Patients Affected by Hemiparesis Due to Cerebrovascular Accident
Brief Title: "Equistasi" and Gait in Hemiparesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Equistasi.01
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- treatment (Experimental): 3 "Equistasi" devices will be placed during physiotherapy, 5 times per week, for 4 weeks
  Interventions: Device: equistasi
- controls (Placebo Comparator): 3 "placebo" devices will be placed during physiotherapy, 5 times per week, for 4 weeks
  Interventions: Device: placebo

INTERVENTIONS:
Device: equistasi — 3 devices will be placed in each patient: 1 at the spinosus process of L5; 1 at the insertion of transverse abdominis; 1 at the insertion of the gluteus medius to the femur. The devices will be kept for 55 minutes, during standard Physiotherapy
  Arms: treatment
Device: placebo — 3 devices will be placed in each patient: 1 at the spinosus process of L5; 1 at the insertion of transverse abdominis; 1 at the insertion of the gluteus medius to the femur. The devices will be kept for 55 minutes, during standard Physiotherapy
  Arms: controls

SUMMARY:
The purpose of the study is to evaluate the effect of "Equistasi" device on quantitative and qualitative gait characteristics in patients affected by hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* subacute hemiparesis
* Functional Ambulation Classification <4

Exclusion Criteria:

* previous neurological deficits
* Glasgow Coma Scale <13
* Complete sensory deficit in the lower limbs
* Levels of Cognitive Functioning ≤5
* polyneuropathy
* contraindications to mobilization/verticalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disability change assessed using Functional Independence Measure scale | 0. 30. 60. 120 days
balance change assessed using Berg Balance Scale | 0. 30. 60. 120 days
gait pattern change assessed using Functional Ambulation Classification scale | 0. 30. 60. 120 days
gait speed change assessed using Timed Up and Go scale | 0. 30. 60. 120 days
gait pattern change using Tinetti scale for gait | 0. 30. 60. 120 days
gait speed change assessed using 10 meter walking test scale | 0. 30. 60. 120 days
swaying of the center of gravity change assessed with stabilometric platform indexes | 0. 30. 60. 120 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Brain Injury and Parkinson Disease Rehabilitation, "Moriggia-Pelascini" Hospital, Gravedona, CO, Italy